CLINICAL TRIAL: NCT06077279
Title: Effect of Horticultural Therapy Program on Psychological Wellbeing, Hope, and Social Adjustment Among Patients With Psychotic Disorders
Brief Title: HCT Effect Among Patients With Psychotic Disorders
Acronym: HCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00013620(9/19/2025)
Record Dates: First submitted 2023-08-29; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Psychotic Disorders
Keywords: Hope; Psychological Adjustment; Psychological Wellbeing; Horticulture Therapy
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horticultural Therapy (Experimental): receive horticulture therapy by seven sessions within two months
  Interventions: Behavioral: Horticultural Therapy Program
- Routine hospital care (No Intervention): doesn't receive horticulture therapy but receive routine care by hospital within conducting the research

INTERVENTIONS:
Behavioral: Horticultural Therapy Program — Horticultural Therapy Program Is selected plant therapy
  Arms: Horticultural Therapy

SUMMARY:
Horticulture therapy has been found to have positive effects on individuals with psychotic disorders, promoting social interaction, reducing social isolation, and improving cognitive function. Effectiveness of horticulture therapy in enhancing well-being, reducing symptoms, and facilitating social adjustment in this population

DETAILED DESCRIPTION:
Horticulture therapy involves gardening and plant-related activities as a form of therapeutic intervention, enhance patient to be mindful to current environment and promote relaxation which can reduce symptoms such as anxiety, depression, and social isolation, improve cognitive function, and promote overall well-being .With this respect, there is an urgent need to find a sustainable and eco-friendly solution for this complex issue by returned to nature and utilizing the low cost and current resources at the same time to make a signification reduction in the psychotic disorder's symptoms

ELIGIBILITY:
Inclusion and exclusionCriteria:

did not undergo any other intervention during the HT program used in the study, just routine care in hospital -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Effect of Horticultural Therapy Program on hope level among patients with psychotic disorders | three months
  Effect of Horticultural Therapy Program may enhance hope by Herth Hope Index among patients with psychotic disorders as Herth Hope Index score ranged from 12 to 48, with higher score indicated higher hope.
Effect of Horticultural Therapy Program on psychological wellbeing level among patients with psychotic | three months
  Effect of Horticultural Therapy Program may enhance psychological wellbeing by Ryff psychological wellbeing scale among patients with psychotic disorders a Ryff psychological wellbeing scale score ranged from 18 to 126 with Higher scores mean higher levels of psychological well-being.
Effect of Horticultural Therapy Program on social adjustment level among patients with psychotic | three month
  Effect of Horticultural Therapy Program may enhance social adjustment by The Modified Social Adjustment Score ranged from 45 to 225 with Higher scores mean higher levels of social adjustment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atta MHR, Salama EAA, Menessy RFM. Effect of Horticultural Therapy Program on Psychological Wellbeing, Hope and Social Adjustment Among Patients With Psychotic Disorders: A Nursing Perspective. J Psychiatr Ment Health Nurs. 2025 Oct;32(5):1035-1052. doi: 10.1111/jpm.13180. Epub 2025 Jun 14. PMID 40515548

DOCUMENTS (1):
  • Study Protocol (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT06077279/Prot_000.pdf